CLINICAL TRIAL: NCT06748183
Title: Effects of Functional Power Training on Mobility and Gait Parameters in Children With Cerebral Palsy.
Brief Title: Functional Power Training on Mobility and Gait Parameters in Cerebral Palsy
Acronym: FPTCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/0706
Record Dates: First submitted 2024-11-03; First posted 2024-12-27 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Gait Parameters; Mobility; Functional Power Training
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: It will be a randomized control trial employing nonprobability convenient sampling. Two groups, comprising participants aged 6 to 12, will be formed and randomly divided. Group A will undergo Functional Power Training (FPT) alongside Routine Physical Therapy (RPT), while Group B will receive only Routine Physical Therapy (RPT). This intervention aims to compare the effects of combined functional training and routine therapy against routine therapy alone, focusing on improvements in gait parameters and mobility among children with Cerebral Palsy.
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional Power Training (Experimental): Group A will participate in Functional Power Training (FPT) alongside routine physical therapy for children with Cerebral Palsy. The standard therapy includes hot packs for muscle relaxation, isometric exercises for motor skills, muscle strength, and coordination, as well as passive stretching. Therapists will also utilize sit-to-stand exercises to enhance gait and overall functional abilities. Over a 14-week intervention period, FPT will include three 60-minute sessions each week, focusing on improving walking capacity and muscle strength. Each session will consist of a 10-minute warm-up, 35 minutes of 3 to 4 power exercises, and a 15-minute cool-down phase, conducted in small groups of 3-6 children with a supervising therapist. Participants will wear sports shoes without orthoses, and power exercises will target functional, multi-joint movements, emphasizing ankle push-off and velocity, with adjustments made for progressive challenges.
  Interventions: Other: Functional Power Training
- Routine Physical therapy (Other): Routine physical therapy for children with Cerebral Palsy includes hot packs for muscle relaxation and isometric exercises aimed at improving motor skills, muscle strength, and coordination. Passive stretching is also part of the treatment plan. Therapists use sit-to-stand exercises to enhance gait, posture, and overall functional abilities. Regular progress evaluations are conducted to adjust interventions as needed, ensuring continuous improvement. The overall goal is to optimize mobility, enhance walking ability, and improve the child's quality of life.
  Interventions: Other: Routine physical therapy

INTERVENTIONS:
Other: Functional Power Training — Group A will participate in Functional Power Training (FPT) alongside routine physical therapy The exercise protocol aims to enhance strength, mobility, and endurance through resistance training across various functional activities. It includes exercises such as running, walking, chair pushing, stair climbing, propelling a stable scooter, and sideways walking, all performed at 50-70% of the participant's maximum speed. Resistance is added using methods like dragging a loaded box with a belt during running and walking, pushing a chair with a loaded box underneath, wearing a loaded vest while climbing stairs, and attaching a loaded box to a scooter for propulsion exercises. Each exercise involves 6 to 8 repetitions lasting 25 seconds, followed by 30 to 50 seconds of rest. This structured regimen focuses on controlled movement and endurance, providing a comprehensive approach to improving physical performance.
  Arms: Functional Power Training
Other: Routine physical therapy — Routine physical therapy for a child with Cerebral Palsy involves hot pack for muscle relaxation and isometric exercises to enhance motor skills, muscle strength, and coordination. Passive stretching will be given as a treatment plan. Therapists employ sit to stand exercise to improve gait, posture, and overall functional abilities. Regular progress evaluations are conducted to adjust interventions, ensuring ongoing improvements.
  Arms: Routine Physical therapy

SUMMARY:
Cerebral Palsy is a lifelong neuromuscular disorder impacting movement, posture, and muscle control, ranging from mild hand weakness to severe paralysis. Risk factors are grouped into specific stages: preconception (linked to the mother's health), prenatal (during pregnancy), perinatal (at birth), and the neonatal and infant stages. Functional power training is employed to improve the functional abilities of children with Cerebral Palsy by involving them in various power-based exercises to strengthen muscles, increase power, and build endurance. This study aims to evaluate the impact of functional power training on gait and mobility in children with Cerebral Palsy.

DETAILED DESCRIPTION:
Cerebral Palsy (CP) is a chronic neuromuscular disorder that affects movement, posture, and muscle control, with symptoms ranging from mild weakness to severe paralysis. The risk factors for CP are classified into preconception, prenatal, perinatal, and neonatal categories. Functional power training (FPT) is a therapeutic approach aimed at improving muscle strength, power, and endurance in children with CP. This study seeks to evaluate the impact of FPT on gait parameters and mobility in children with CP. This randomized controlled trial will include 26 children, aged 6 to 12 years, with Gross Motor Function Classification System (GMFCS) I or II. Participants will be randomly assigned to either the experimental group (FPT plus routine physical therapy) or the control group (routine physical therapy alone). Exclusion criteria include recent botulinum toxin A treatment, serial casting within the last 6 months, or selective dorsal rhizotomy. Gait parameters (step length, stride length, cadence, gait speed, and step width) and mobility outcomes (6MWT and Timed Up and Go test) will be assessed before and after the intervention. Data will be analyzed using SPSS version 23.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 to 12
* Gross Motor Function Classification System (GMFCS) I and II
* Either gender will be included

Exclusion Criteria:

* Treatment with botulinum toxin A in lower limb
* Serial Casting of lower limb less than 6 months before the start of the functional power training
* Selective dorsal rhizotomy treatment
* Children who did not (yet) choose walking as their preferred way of mobility

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2024-09-26 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Step length | 5 months
  To measure step length(centimeters), first mark a starting point on the floor, then have the participant walk naturally while measuring the distance between consecutive heel strikes. Repeat this process for several steps and calculate the average of those measurements to determine the participant's typical step length.
Stride length | 5 months
  To measure stride length(meters) first identify the starting point on the walking path and instruct the participant to take several steps. Then, measure the distance between two consecutive heel strikes of the same foot, repeat for multiple strides, and calculate the average to determine the participant's typical stride length.
Cadence | 5 months
  To measure cadence(steps/min), choose a specific time interval and instruct the participant to walk within that period while counting the number of steps taken. Repeat the process for accuracy and calculate the average steps per minute to determine the participant's cadence.
Gate speed | 5 months
  To measure gait speed(meters/sec), mark the starting and finishing points on a straight path, and instruct the participant to walk at a comfortable pace while measuring the time taken to cover the distance. Repeat the process for accuracy, then calculate gait speed by dividing the distance by the time taken to complete it.
Step width | 5 months
  To measure step width(centimeter), define a walking path and instruct the participant to walk naturally while measuring the lateral distance between the midpoints of successive footsteps. Repeat this measurement for multiple steps and calculate the average step width to analyze the participant's walking pattern.

SECONDARY OUTCOMES:
6-Minute Walk Test | 5 months
  Set up a marked straight pathway and instruct the individual to walk as far as possible within a 6-minute timeframe, encouraging them to maintain a consistent pace while providing periodic time updates. At the end of the session, measure the total distance covered in meters to assess their functional capacity
Timed up and go (TUG) test | 5 months
  Start with the individual seated in a chair, and upon the signal, have them stand, walk three meters, turn, walk back, and sit down. Measure the total time taken for this sequence to assess functional mobility, with longer times suggesting potential mobility challenges.

CONTACTS AND LOCATIONS:
Overall Officials: Asiah Fareed, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Vulpen LF, de Groot S, Rameckers E, Becher JG, Dallmeijer AJ. Improved Walking Capacity and Muscle Strength After Functional Power-Training in Young Children With Cerebral Palsy. Neurorehabil Neural Repair. 2017 Sep;31(9):827-841. doi: 10.1177/1545968317723750. Epub 2017 Aug 8. PMID 28786309